CLINICAL TRIAL: NCT04403828
Title: Impact of COVID-19 on Personal Protection Among Dentist in Egypt: A Quick Online Survey
Brief Title: Impact of COVID-19 on Personal Protection Among Dentist in Egypt
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Other Study IDs: PPE in COVID-19
Record Dates: First submitted 2020-05-24; First posted 2020-05-27 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: COVID 19
Keywords: COVID-19; Personal Protection; Dentist; Egypt
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — a cross-sectional, online survey-based study administered to Dentist in Egypt. A 20-item questionnaire developed and distributed using Google Forms.

SUMMARY:
Dentist exposed to coronavirus (COVID-19) may not have adequate access to personal protective equipment (PPE), safety procedures, and diagnostic protocols. Our objective will be to evaluate the reality and perceptions about personal safety among dentist in Egypt

DETAILED DESCRIPTION:
This is a cross-sectional, online survey-based study administered to Dentist in Egypt. A 20-item questionnaire will be developed and distributed using Google Forms.

Participants were recruited through social networking websites and applications (Twitter, Instagram, Facebook, LinkedIn, and WhatsApp). The questionnaire will be conducted from 24 May 2020 and until 30 june 2020.

The survey will be delivered in Enlish. Participants will be able to complete the survey only once and will be allowed to terminate the survey at any time they desired. The survey will be anonymous and confidential. An introductory paragraph outlining the purpose of the study will be posted along with the survey.

ELIGIBILITY:
Inclusion Criteria:

All dentist actively working in Egypt

Exclusion Criteria:

* non dentist
* resident outside egypt

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dentist
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Personal protection measures | one week
  measure the personal protection measures used among dentist during Covid-19 pandemic through online Survey

SECONDARY OUTCOMES:
impact of Covid-19 pandemic on type of face masks used in dental clinic | one week
  measure the personal protection measures used among dentist during Covid-19 pandemic through online Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Odeh ND, Babkair H, Abu-Hammad S, Borzangy S, Abu-Hammad A, Abu-Hammad O. COVID-19: Present and Future Challenges for Dental Practice. Int J Environ Res Public Health. 2020 Apr 30;17(9):3151. doi: 10.3390/ijerph17093151. PMID 32366034
- [Background] Ather A, Patel B, Ruparel NB, Diogenes A, Hargreaves KM. Coronavirus Disease 19 (COVID-19): Implications for Clinical Dental Care. J Endod. 2020 May;46(5):584-595. doi: 10.1016/j.joen.2020.03.008. Epub 2020 Apr 6. PMID 32273156
- [Background] Alharbi A, Alharbi S, Alqaidi S. Guidelines for dental care provision during the COVID-19 pandemic. Saudi Dent J. 2020 May;32(4):181-186. doi: 10.1016/j.sdentj.2020.04.001. Epub 2020 Apr 7. PMID 32292260